CLINICAL TRIAL: NCT05584124
Title: Neuromodulation for Rehabilitation of Post-Stroke Fatigue: An rTMS Pilot Study
Brief Title: rTMS for Post-stroke Fatigue
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI is transfering from Charleston SC to Atlanta GA. The trial will resume once the PI completes his transfer. Modifications will be made to the trial once the ethical/regulatory approvals are recieved from the new station.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Ralph H. Johnson VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N3790-W; IK2RX003790 (NIH); 00120805 (Other: Ralph H. Johnson VA Medical Center)
Record Dates: First submitted 2022-10-07; First posted 2022-10-18 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Stroke; Stroke, Chronic; Fatigue
Keywords: non-invasive brain stimulation; post-stroke fatigue; perception of fatigue; repetitive transcranial magnetic stimulation; rTMS
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome; Fatigue

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to their groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Real M1 High Frequency rTMS (Experimental): Participants will be randomly assigned to receive high-frequency repetitive transcranial magnetic stimulation (rTMS) to the top of their head for approximately 40 minutes.
  Interventions: Device: High frequency repetitive transcranial magnetic stimulation
- Real LDLPFC High Frequency rTMS (Experimental): Participants will be randomly assigned to receive high-frequency repetitive transcranial magnetic stimulation (rTMS) to the left frontal part of their head for approximately 40 minutes.
  Interventions: Device: High frequency repetitive transcranial magnetic stimulation
- Sham rTMS (Sham Comparator): Participants will be randomly assigned to receive sham/placebo repetitive transcranial magnetic stimulation (rTMS) to the their head for approximately 40 minutes. This is a control condition.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: High frequency repetitive transcranial magnetic stimulation — MAGSTIM Super Rapid2 Plus
  Arms: Real LDLPFC High Frequency rTMS; Real M1 High Frequency rTMS
Device: Sham repetitive transcranial magnetic stimulation — MAGSTIM Super Rapid2 Plus
  Arms: Sham rTMS

SUMMARY:
This experimental trial is investigating the use of magnetic stimulation of the brain as a possible treatment for people with post-stroke fatigue. Fatigue is a common condition after a stroke and can negatively impact an individual's ability to perform desired social and physical activities. Magnetic stimulation of the brain has been shown to improve signs and symptoms of related psychological (e.g., depression) conditions. Participants in this trial will receive a type of magnetic stimulation called repetitive magnetic stimulation, or rTMS. The investigators will measure feelings of fatigue, and other clinical characteristics related to mood and cognition, before and after participants receive rTMS.

ELIGIBILITY:
Inclusion Criteria:

* 35 - 80 years of age
* more than 6 months post-stroke
* able to walk 10m unassisted
* Clinically present fatigue

Exclusion Criteria:

* Contraindications to MRI/TMS/rTMS (e.g. implanted metal within the head, history of seizures)
* Inability to follow simple three-step instructions
* Multiple strokes on opposite hemispheres
* Cerebellar and/or brainstem strokes
* Diagnosed comorbid neurological conditions (e.g. multiple sclerosis, Parkinson's disease, moderate/severe TBI)
* Comorbid psychological conditions (e.g. depression, anxiety, PTSD)
* strokes within stimulation sites
* Pregnancy
* Severe hypertension (resting SBP > 200, DBP > 120)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2027-10-29 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Change in Fatigue Severity Scale (FSS) score | Change from baseline FSS score to 7 days after last treatment
  The Fatigue Severity Scale (FSS) is a patient reported outcome measure assessing perceived influence of fatigue over the past week. The scale consists of nine questions measured on a 7-point Likert scale (1-7). The FSS' range of scores is from 9 (min) to 63 (max) with lower numbers representing lower/less impact of fatigue.

SECONDARY OUTCOMES:
Change in Modified Fatigue Impact Scale (MFIS) score | Change from baseline MFIS score to 7 Days after last treatment
  The Modified Fatigue Impact Scale (MFIS) is a Patient reported outcome assessing the impact of fatigue over the past four weeks. The questionnaire is comprised of 21 questions covering three domains (physical, cognitive, and psychosocial subscales). The assessment is graded on a 5 point Likert scale (0-4). The MFIS' range of scores is from 0-84 with higher scores indicating greater impact/worse fatigue. The range of scores for the physical, cognitive, and psychosocial subscales are 0-36, 0-40, and 0-8 respectively. Greater scores indicate greater/worse impact of fatigue.
Change in Fatigue Severity Scale (FSS) score | Change from baseline FSS score to 3 months after last treatment
  The Fatigue Severity Scale (FSS) is a patient reported outcome measure assessing perceived influence of fatigue over the past week. The scale consists of nine questions measured on a 7-point Likert scale (1-7). The FSS' range of scores is from 9 (min) to 63 (max) with lower numbers representing lower/less impact of fatigue.
Change in Modified Fatigue Impact Scale (MFIS) score | Change from baseline MFIS score to 3 months after last treatment
  The Modified Fatigue Impact Scale (MFIS) is a Patient reported outcome assessing the impact of fatigue over the past four weeks. The questionnaire is comprised of 21 questions covering three domains (physical, cognitive, and psychosocial subscales). The assessment is graded on a 5 point Likert scale (0-4). The MFIS' range of scores is from 0-84 with higher scores indicating greater impact/worse fatigue. The range of scores for the physical, cognitive, and psychosocial subscales are 0-36, 0-40, and 0-8 respectively. Greater scores indicate greater/worse impact of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: John H Kindred, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No